CLINICAL TRIAL: NCT05964621
Title: Venous Thromboembolism in Patients Undergoing Primary Pancreatic Tumour Resection; a Prospective Observational Study
Brief Title: Venous Thromboembolism in Primary Pancreatic Tumour Resection
Acronym: PaTR-VTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anaesthesiology, University of Thessaly
Other Study IDs: 24165
Record Dates: First submitted 2023-07-03; First posted 2023-07-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Venous Thromboembolism; Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Venous Thromboembolism; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreatic cancer patients undergoing pancreatic cancer resection: Perioperative laboratory examinations will follow institutional guidelines. These will include, but will not be limited to full blood count, conventional coagulation tests, liver function, and kidney function tests. Moreover, for the purpose of this study, the following parameters will also be obtained; vWF, factors VIII and XI, D-dimers, fibrinogen, platelets activation (multiplate), adams-13, anti-Xa and high sensitivity troponin. All samples will be obtained via puncture from a peripheral vein. Blood samples will obtained at three time points; preoperatively before induction to GA (01), early postoperatively in PACU (02) and postoperatively before discharge (10 days, 03). Of note, at 30 days our patients will undergo an evaluation for asymptomatic DVT with a US triplex scanner. In addition, any thromboembolic episode (deep vein thrombosis, pulmonary embolism) will also be recorded.

SUMMARY:
This study will evaluate the development of venous thromboembolism (VTE) and possible determinants in patients with primary pancreatic cancer undergoing pancreatic cancer resection.

DETAILED DESCRIPTION:
Cancer associated thrombosis (CAT) is the second cause of death, in oncologic patients after tumour progression itself. Patients suffering from malignancies are at increased risk for both venous (4-20%) and arterial (2-5%) thrombotic events. Moreover, cancer is one of the most important acquired risk factors for the development of venous thromboembolism (VTE).

Pancreatic cancer is the fourth most deadly cancer world-widely and has been recognised as the most prothrombotic malignancy, with a reported incidence of VTE (8-18%), followed by renal and ovarian cancer (VTE 5.6%). Although the exact pathophysiological mechanisms are still poorly understood it seems that pancreatic cancer induces a prothrombotic and hypercoagulable state.

Aims

* To evaluate the predictive value of preoperatively or early postoperatively obtained NLR, in patients with primary pancreatic cancer undergoing pancreatic cancer resection, for VTE up to the 30rd postoperative day
* To evaluate the predictive value of preoperatively or early postoperatively obtained coagulation biomarkers/parameters, in patients with primary pancreatic cancer undergoing pancreatic cancer resection, for VTE up to the 30rd postoperative day
* To evaluate the incidence of VTE in patients with primary pancreatic cancer undergoing pancreatic cancer resection
* To assess the perioperative coagulation status of patients with primary pancreatic cancer undergoing pancreatic cancer resection
* To evaluate any possible determinant or predictive factor for VTE among the coagulation parameters or patients' baseline characteristics

ELIGIBILITY:
Inclusion Criteria:

* Consecutive pancreatic cancer patients undergoing pancreatic cancer resection in University Hospital of Larissa, after informed consent will be included.

Exclusion Criteria:

* Refuse to participate
* Previous thromboembolic event < 6 months prior to the operation
* History of inherited or acquired bleeding disorder
* ASA PS > 3
* Concomitant presence of a second primary malignancy
* Unresectable pancreatic cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary pancreatic cancer are appropriately staged with high quality imaging according to the NCCN guidelines version 1.2023. Surgical resection is the only potentially curative technique for the management of pancreatic cancer. However, the median survival even of patients submitted to resection remains low, ranging between 15 and 19 months.
  The negative margin status is probably the most important prognostic factor. Pancreatic tumours are classified as resectable, borderline resectable and unresectable based on the probability of attaining an R0 resection.In borderline resectable neoadjuvant chemotherapy is administered in these patients prior to resection. In regards to the Whipple's procedure, the aim is to preserve the pylorous while, performing a pancreaticojejunostomy for the reestablishment of the gastrointestinal tract continuity.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Neutrophil to lymphocyte ratio-VTE | up to 30rd postoperative day
  The predictive value of preoperatively or early (10th day) postoperatively obtained neutrophil to lymphocyte ratio (NLR), in patients with primary pancreatic cancer undergoing pancreatic cancer resection, for VTE up to the 30rd postoperative day
von Willebrand factor-VTE | up to 30rd postoperative day
  The predictive value of preoperatively or early (10th day) postoperatively obtained von Willebrand factor in patients with primary pancreatic cancer undergoing pancreatic cancer resection, for VTE up to the 30rd postoperative day
Factors VIII and XI-VTE | up to 30rd postoperative day
  The predictive value of preoperatively or early (10th day) postoperatively obtained factors VIII and XI in patients with primary pancreatic cancer undergoing pancreatic cancer resection, for VTE up to the 30rd postoperative day
D-dimers-VTE | up to 30rd postoperative day
  The predictive value of preoperatively or early (10th day) postoperatively obtained, D-dimers, in patients with primary pancreatic cancer undergoing pancreatic cancer resection, for VTE up to the 30rd postoperative day
Fibrinogen-VTE | up to 30rd postoperative day
  The predictive value of preoperatively or early (10th day) postoperatively obtained, fibrinogen, in patients with primary pancreatic cancer undergoing pancreatic cancer resection, for VTE up to the 30rd postoperative day
Adams-13-VTE | up to 30rd postoperative day
  The predictive value of preoperatively or early (10th day) postoperatively obtained adams-13 in patients with primary pancreatic cancer undergoing pancreatic cancer resection, for VTE up to the 30rd postoperative day
VTE incidence in primary pancreatic cancer resection | up to 30rd postoperative day
  The incidence of VTE in patients with primary pancreatic cancer undergoing pancreatic cancer resection

CONTACTS AND LOCATIONS:
Overall Officials: Eleni M Arnaoutoglou, Professor, Study Chair — Dpt of Anaesthesiology; Dimitrios Zacharoulis, Professor, Principal Investigator — Dpt of Surgery; Paraskevi Kotsi, Asst Professor, Principal Investigator — Dpt of Transfusion Medicine; Dimitrios Symeonidis, Asst Professor, Principal Investigator — Dpt of Surgery; Maria P Ntalouka, M.D., Ph.D, M.Sc., Principal Investigator — Dpt of Anaesthesiology
Locations (1):
- University Hospital of Larissa, Larissa, Thessaly, Greece

REFERENCES:
- [Derived] Ntalouka MP, Symeonidis D, Kotsi P, Petinaki E, Matsagkas M, Tepetes K, Zacharoulis D, Arnaoutoglou EM. Venous thromboembolism in patients undergoing pancreatic cancer surgery (PaTR-VTE) with curative intent; protocol of a prospective observational study. BMC Surg. 2025 Apr 26;25(1):183. doi: 10.1186/s12893-024-02665-z. PMID 40287701